CLINICAL TRIAL: NCT07116200
Title: Effectiveness of an Early Reading Intervention for Young Children With Intellectual Disabilities Who Need or Use Augmentative and Alternative Communication: A Randomized Controlled Trial
Brief Title: Effectiveness of an Early Reading Intervention for Young Children With Intellectual Disabilities Who Need or Use Augmentative and Alternative Communication
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold University College (Other)
Collaborators: University of Oslo (Other); University of South-Eastern Norway (Other); Karolinska Institutet (Other); Heidelberg University (Other); Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NRC: 353017
Record Dates: First submitted 2025-06-20; First posted 2025-08-11 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Education
Keywords: Literacy intervention; Intellectual disability; Augmentative and alternative communication (AAC); Phonological awareness; Phonemic awareness; Early intervention; Special education; Kindergarten-based intervention; School-based intervention; Reading development
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Combined Intervention: Kindergarten and First Grade (Experimental): Participants in this arm will receive a structured literacy intervention in both kindergarten and first grade. The kindergarten intervention focuses on developing early literacy skills, including phonological awareness and phonemic awareness. In first grade, the intervention builds on these foundational skills and targets more advanced reading abilities, such as decoding and sight word recognition. Individualized intervention sessions are delivered by the participant's designated special needs educator or teacher at their respective kindergarten or school. This arm is designed to assess the cumulative effects of receiving both early literacy and reading interventions across kindergarten and first grade.
  Interventions: Other: Early Literacy Intervention in Kindergarten; Other: Literacy Intervention in First Grade
- Intervention in Kindergarten and Training as Usual in First Grade (Experimental): Participants in this arm will receive a structured literacy intervention in kindergarten and training as usual in first grade. The kindergarten intervention focuses on developing early literacy skills, including phonological awareness and phonemic awareness. In first grade, participants will receive training as usual, meaning they will follow the standard school curriculum without additional literacy intervention from the study. This arm is designed to evaluate the effects of early intervention alone, without follow-up support in first grade.
  Interventions: Other: Early Literacy Intervention in Kindergarten
- Training as Usual in Kindergarten and Reading Intervention in First Grade (Experimental): Participants in this arm will receive training as usual during kindergarten and a structured reading intervention in first grade. During kindergarten, they will attend regular classroom instruction without receiving any early literacy intervention from the study. In first grade, they will participate in individualized reading intervention sessions focused on early literacy skills, decoding and sight word recognition, delivered by trained educators or specialists. This arm is designed to evaluate the effects of the first-grade reading intervention alone, without prior early literacy support.
  Interventions: Other: Literacy Intervention in First Grade
- Training as Usual in Kindergarten and First Grade (No Intervention): Participants in this arm will receive training as usual during both kindergarten and first grade. They will attend standard classroom instruction without receiving any additional literacy intervention from the study. This arm serves as the control group and is designed to evaluate typical developmental progress in the absence of targeted intervention.

INTERVENTIONS:
Other: Early Literacy Intervention in Kindergarten — In the kindergarten intervention, children will receive early literacy instruction through the Early Literacy Program, adapted for those using augmentative and alternative communication. Based on Accessible Literacy Learning by Light and McNaughton, the program enables nonverbal responses such as signs, symbol pointing, or eye-gaze, removing the need for speech. Instruction follows evidence-based practices including direct and explicit teaching, scaffolding, immediate feedback, cumulative review, practice, and subvocal rehearsal. The program targets five foundational literacy skills: phonological awareness, letter-sound correspondence, sound blending, shared reading, and understanding concepts about print. Supplementary materials such as flashcards and lotto games will also be used to reinforce learning.
  Arms: Combined Intervention: Kindergarten and First Grade; Intervention in Kindergarten and Training as Usual in First Grade
Other: Literacy Intervention in First Grade — In the first-grade intervention, students will receive literacy instruction using the Reading for All program, which is adapted for children who use augmentative and alternative communication. Based on Accessible Literacy Learning by Light and McNaughton, the program allows responses through nonverbal methods like signs, symbol pointing, or eye-gaze, eliminating the need for oral replies. Instruction is grounded in evidence-based practices such as direct and explicit instruction, scaffolding, immediate corrective feedback, cumulative review, practice, and subvocal rehearsal. Reading for All addresses six key literacy skills: sound blending, letter-sound correspondence, phoneme segmentation, sight word recognition, shared reading, and decoding. Additional activities (flashcards and lotto games) will be a supplement to the material.
  Arms: Combined Intervention: Kindergarten and First Grade; Training as Usual in Kindergarten and Reading Intervention in First Grade

SUMMARY:
The goal of this 2x2 factorial randomized controlled trial is to evaluate the effectiveness of two literacy interventions delivered at different time points, in kindergarten and in first grade, on the development of literacy skills in children with intellectual disabilities who require augmentative and alternative communication. The main questions it aims to answer are:

* Does early intervention in kindergarten lead to greater improvements in phonological and phonemic awareness, vocabulary, and articulation compared to training as usual?
* Does a follow-up intervention in first grade enhance decoding skills and sight word recognition beyond the gains achieved through the kindergarten intervention alone?
* Does phonological awareness at the end of kindergarten mediate the relationship between early intervention and later outcomes in vocabulary, articulation, and decoding?
* Do children who receive both interventions perform better than those who receive only one or none (training as usual), suggesting a cumulative or higher-dose effect?

Researchers will compare four arms formed through a 2x2 factorial design after randomization to see if whether timing, combination, and sequencing of interventions produce differential effects on literacy outcomes.

Participants will:

* In kindergarten receive either an early literacy intervention or training as usual.
* In first grade receive either a follow-up literacy intervention or training as usual, depending on group allocation.
* Be assessed at key time points in both years, measuring phonological awareness, phonemic awareness, vocabulary, and articulation in kindergarten, and expanding to include decoding and sight word recognition in first grade.

DETAILED DESCRIPTION:
Literacy skills are fundamental in modern society. A significant portion of information is conveyed through written language. With the widespread use of the internet, written communication has become even more influential in our daily lives. The ability to read and write supports cognitive development, enhances social interactions, improves comprehension, and contributes to academic achievement. Conversely, a lack of literacy skills can limit access to general knowledge and deprive individuals of these important benefits.

One group that stands to gain significantly from literacy skills is individuals with intellectual disabilities who use augmentative and alternative communication. For these individuals, reading and writing can lead to enhanced self-esteem and increased opportunities for inclusion in school, the workplace, and the broader community.

Research has shown that individuals with intellectual disabilities who use augmentative and alternative communication can learn to read and write. However, it is crucial that literacy instruction is tailored to their specific needs.

ELIGIBILITY:
Inclusion Criteria:

* children diagnosed with intellectual disability, confirmed by multidisciplinary assessments carried out by the Child rehabilitations service or currently undergoing such an evaluation
* ages 4-8 (the last year in kindergarten)
* lack of functional speech and must use augmentative and alternative communication as the primary form of communication
* have a (designated) special education kindergarten teacher

Exclusion Criteria:

* having a severe visual or hearing impairment
* children who can decode syllables or words
* children with severe physical disabilities prevent the children from being able to answer with their fingers, unless they can respond with eye pointing or signs

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Phonological Awareness and Letter-Sound Correspondence Assessed in Kindergarten | 5 weeks
  All participants will be assessed five times in phonological awareness and letter-sound correspondence during their final year of kindergarten. These tests are part of the Reading for All materials.
Phonological Awareness, Letter-Sound Correspondence and Decoding Assessed in First Grade | 5 weeks
  All participants will be assessed five times in phonological awareness, letter-sound correspondence and decoding during first grade. These tests are part of the Reading for All materials.

SECONDARY OUTCOMES:
Vocabular assessment in kindergarten | 2 weeks
  All participants will be assessed twice using the MacArthur-Bates Communicative Development Inventories before and after the kindergarten intervention.
Vocabular assessment in first grade | 1 week
  All participants will be assessed using the MacArthur-Bates Communicative Development Inventories after the first grade intervention.
Articulation assessment in kindergarten | 2 weeks
  All participants will be assessed before and after the kindergarten intervention.
Articulation assessment in first grade | 1 week
  All participants will be assessed after the first grade intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Nordahl-Hansen, PhD, Principal Investigator — Østfold University College
Locations (1):
- Østfold University College, Halden, Østfold fylke, Norway

IPD SHARING:
Plan to Share IPD: Yes
Following the Findable, Accessible, Interoperable, Reusable Data Principles, the trial protocol, its registration, and models created to analyse the data during the project will be made available on platforms such as Open Science Framework and https://clinicaltrials.gov/. Project objectives and results will be communicated to the general public through newsletters, social media, mainstream media (regional newspaper), and presentations at showcase events. Lastly, we plan to launch a publicly accessible website of the project, describing the project, including its goals and the partners.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Study protocol: August 2025- August 2028 Statistical analysis Plan: August 2026- December 2027 Analytic Code: August 2026- December 2027